CLINICAL TRIAL: NCT01581749
Title: Prospective Evaluation of Truebeam STX Stereotactic Body Radiosurgery for Low and Intermediate Risk Prostate Cancer
Brief Title: Evaluation of Truebeam for Low-Intermediate Risk Prostate Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Albert DeNittis (Other)
Responsible Party: Sponsor-Investigator, Albert DeNittis, Chief, Radiation Oncology. Lankenau Medical Center, Main Line Health, Main Line Health
Organization: Main Line Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R12-3104L
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Prostate Neoplasms
Keywords: low risk prostate cancer; intermediate risk prostate cancer; stereotactic radiosurgery
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 36.25Gy to prostate in 5 fractions (Other): 36.25Gy to be delivered to the prostate in 5 fractions. There is only 1 arm in this study.
  Interventions: Radiation: "TrueBeam" stereotactic body radiosurgery

INTERVENTIONS:
Radiation: "TrueBeam" stereotactic body radiosurgery — 36.25Gy to be delivered to the prostate in 5 fractions. There is only 1 arm in this study.

SUMMARY:
The primary safety purpose of this study is to estimate the rates of immediate and long-term high grade (grade 3-5) gastrointestinal and genitourinary side effects during the five years after TrueBeam stereotactic body radiotherapy in low-risk and intermediate-risk prostate cancer patients. The primary efficacy purpose is to compare 5 year biochemical disease free survival rates with TrueBeam to 5 year biochemical diseases free survival rates with dose-escalated external beam radiation therapy.

DETAILED DESCRIPTION:
The prescribed PTV dose of 36.25Gy shall be given in 5 fractions using the Truebeam STx.

At one week after treatment, toxicity and AUA score will be evaluated. At 1 month following treatment, patients will be assessed for acute toxicity, and will fill out AUA form, SF-12, EPIC-26, SHIM and Utilization of Sexual Rx/Devices. At 3, 6, 12, 18, and 24 month intervals (and every 6 months thereafter, through year 5, and annually through year 10, if investigators opt to continue past year 5), patients will be seen and evaluated, including a history, physical exam, ECOG performance status, PSA, toxicity evaluation, and AUA score. In addition, at 6 months, 12 months and annually thereafter, the SF-12, EPIC-26, SHIM and Utilization of Sexual Medications/Devices will be administered. Examination and studies may be done at outside facility.

A prostate biopsy will be performed at time of biochemical or local clinical failure, and is encouraged at 2 years following treatment and at time of distant failure.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven prostate adenocarcinoma within 1 year of enrollment
* Low risk: Gleason <or=6 & PSA <or=10 & Clinical Stage T1b-T2a,Nx or N0, Mx or M0
* Intermediate risk:Gleason <or=6 & PSA<or=10 & Clinical Stage T2b OR Gleason=7 & PSA<or=10 & Clinical Stage T1b-T2b OR Gleason <or=6 & PSA > 10 & < or =20 & Clinical Stage T1b- T2b, Nx or NO, Mx or M0
* ECOG Performance Status 0-1
* No prior prostate radiation or other definitive therapy

Exclusion Criteria:

* implanted hardware or other material that would prohibit treatment planning or delivery
* chemotherapy for a malignancy within the previous 5 years
* history of an invasive malignancy (other than this prostate cancer,or basal or squamous skin cancers) within prior 5 years
* hormone ablation for 2 months prior to treatment or during treatment

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-10; Primary Completion 2017-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
acute and late GI/GU toxicity rate following treatment | 5 years
  The study is designed to test the null hypothesis that the acute and late GI/GU toxicity rate 5 years following treatment is greater than 10% versus the alternative hypothesis that the toxicity rate is less than or equal to 10%. The sample size is determined such that there is 90% probability, or power, of identifying excessive toxicity if the true toxicity rate is 20% at the one-sided 5% significance level.

SECONDARY OUTCOMES:
a comparison of biochemical disease free survival in low risk patients treated with TrueBeam compared to (historical) biochemical disease free survival in patients treated with dose-escalated external beam radiation therapy | 5 years
  For the low-risk cohort, the study is powered to compare 5-year bDFS rates observed with TrueBeam STx to 5-year bDFS rates reported with dose-escalated external beam RT. In Beaumont's monotherapy HDR series treating LR patients, 5-yr ASTRO bDFS was 98%; in Demanes' series of 75% LR and 25% IR, this was 96%. Since TB delivers doses similar to HDR monotherapy, a conservative estimate of the success rate for TB is 97.5% for LR patients.

CONTACTS AND LOCATIONS:
Overall Officials: Albert DeNittis, MD, Principal Investigator — Lankenau Medical Center, Main Line Health
Locations (1):
- Lankenau Medical Center, Radiation Oncology, Wynnewood, Pennsylvania, United States

REFERENCES:
- [Background] King CR, Lehmann J, Adler JR, Hai J. CyberKnife radiotherapy for localized prostate cancer: rationale and technical feasibility. Technol Cancer Res Treat. 2003 Feb;2(1):25-30. doi: 10.1177/153303460300200104. PMID 12625751